CLINICAL TRIAL: NCT02955667
Title: The Application of Invivo Microscopy Imaging in the Early Diagnosis of Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Fang Li
Record Dates: First submitted 2016-10-29; First posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-10

CONDITIONS: Cervical Cancer; Cervical Precancer
Keywords: invivo microscopy; colposcopy; cervical precancer and cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- invivo microscopy group (Experimental): patients receive invivo micro-colposcopy examination and do not have to receive the biopsies
  Interventions: Procedure: invivo microscopy group
- normal group (Other): patients receive normal colposcopy examination and the biopsy specimens are sent for pathological HE staining and analysis
  Interventions: Procedure: normal group

INTERVENTIONS:
Procedure: invivo microscopy group — patients receive invivo micro-colposcopy examination
  Arms: invivo microscopy group
Procedure: normal group — patients receive normal colposcopy examination and the biopsy specimens are sent for pathological HE staining and analysis
  Arms: normal group

SUMMARY:
This study intends to carry out a prospective, randomized controlled trial to research and development a new invivo microscopy based on the technology which is combined with high-definition microscopy and colposcopy，so as to diagnose cervical lesion directly and non-invasively by observing cervical tissues and cells, which makes it possible to diagnose cervical cancer without wounds.

ELIGIBILITY:
Inclusion Criteria:

1. cervical cytologic test result is HSIL
2. persistent infection with high-risk HPV
3. cervical pathological diagnosis is LSIL or HSIL

Exclusion Criteria:

1. acute infection of lower genital tract
2. the wound in lower genital tract
3. active bleeding in lower genital tract

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy rate | 1 day (time of the examination)

SECONDARY OUTCOMES:
image accordance rate | 1 day (time of the examination)

IPD SHARING:
Plan to Share IPD: No